CLINICAL TRIAL: NCT03006341
Title: Validation of Predictors for Oral Anticoagulant Medication Choice Using EMR Data
Brief Title: Validation of Predictors of OAC Initiation Using EMR Data
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0219
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; Telmisartan; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dabigatran etexilate: NVAF patients initiating dabigatran etexilate
  Interventions: Drug: Dabigatran etexilate
- Warfarin: NVAF patients initiating warfarin
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran etexilate — observed upto 12 months
  Other Names: MICARDIS, PRITOR, TELMISARTAN
  Groups: Dabigatran etexilate
Drug: Warfarin — Observed upto 12 months
  Groups: Warfarin

SUMMARY:
The objectives of this study are, first, to identify select clinical covariates from electronic medical records (EMR) that might be associated with initiation of oral anticoagulant medications (dabigatran or warfarin) in patients with non-valvular atrial fibrillation (NVAF) at risk for stroke; second, to quantify the association between EMR-based clinical characteristics and patterns of insurance claims; third, to assess the potential for unmeasured confounding in dabigatran vs warfarin comparative effectiveness and safety studies based on administrative claims databases.

ELIGIBILITY:
Inclusion Criteria:

* First dispensing of warfarin or dabigatran between October 2010 and December 2014
* Diagnosis of atrial fibrillation
* ≥ 12 months enrolment in the database preceding the date of the first dispensing
* Age ≥ 18
* Congestive Heart Failure, Hypertension, Age > 75, Diabetes Mellitus, Prior Stroke or Transient Ischemic Attack, Vascular Disease (CHA2DS2-VASc) score ≥ 1

Exclusion Criteria:

* Prior use of oral anticoagulation
* Evidence of valvular atrial fibrillation
* Missing or ambiguous age or sex information
* Patients with a nursing home stay during baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a recorded diagnosis of atrial fibrillation without evidence of valvular etiology and at risk for stroke
Sampling Method: Non-Probability Sample
Enrollment: 140187 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A validation study; Patients from a United States health insurance database (linked to electronic medical records (EMR) in a subset) with a recorded diagnosis of atrial fibrillation without evidence of valvular aetiology and at risk for stroke who initiate dabigatran or warfarin between October 2010 and December 2014.
Pre-assignment Details: In this non-interventional study based on existing data, no patients were screened.
Groups:
- Dabigatran Etexilate: Patients from a United States health insurance database (linked to electronic medical records (EMR) in a subset) with a recorded diagnosis of atrial fibrillation without evidence of valvular aetiology and at risk for stroke who initiate dabigatran etexilate between October 2010 and December 2014.
- Warfarin: Patients from a United States health insurance database (linked to electronic medical records (EMR) in a subset) with a recorded diagnosis of atrial fibrillation without evidence of valvular aetiology and at risk for stroke who initiate warfarin between October 2010 and December 2014.
- Rivaroxaban: (Post hoc analysis) Patients from a United States health insurance database (linked to electronic medical records (EMR) in a subset) with a recorded diagnosis of atrial fibrillation without evidence of valvular aetiology and at risk for stroke who initiate rivaroxaban between October 2010 and December 2014.
- Apixaban: (Post hoc analysis) Patients from a United States health insurance database (linked to electronic medical records (EMR) in a subset) with a recorded diagnosis of atrial fibrillation without evidence of valvular aetiology and at risk for stroke who initiate apixaban between October 2010 and December 2014.
Period: Overall Study
Arm/Group | Dabigatran Etexilate | Warfarin | Rivaroxaban | Apixaban
Started (Eligible in the claims database) | 26199 | 70071 | 32595 | 11322
Completed (Successfully linked in the EMR but not necessarily propensity score matched) | 1130 | 2566 | 1602 | 637
Not Completed | 25069 | 67505 | 30993 | 10685
Not completed — Not linked in the EMR | 25069 | 67505 | 30993 | 10685

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are based on all patients who successfully linked in the EMR
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate | Warfarin | Rivaroxaban | Apixaban | Total
Number analyzed (Participants) | 1130 | 2566 | 1602 | 637 | 5935
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: Baseline characteristics are based on all patients who successfully linked in the EMR
  Years | 65.1 (11.4) | 69.3 (11.3) | 66.2 (11.1) | 67.3 (11.4) | 67.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: Baseline characteristics are based on all patients who successfully linked in the EMR
  Participants
    Female | 432 | 1006 | 600 | 250 | 2288
    Male | 698 | 1560 | 1002 | 387 | 3647
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Obesity
Description: Percentage of patients with obesity; where obesity is defined as "obese, not-obese based on note of obesity or recorded body mass index (BMI) > 30 in the electronic medical records (EMR)". The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: Two sets of results are provided, before and after PS matching. Rivaroxaban and Apixaban correspond to post-hoc analyses not pre-specified in the protocol and hence not included in the outcome measures.
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching: number analyzed (Participants) | 857 | 1983
  Before PS matching | 58.2 | 51.7
  After PS matching: number analyzed (Participants) | 641 | 659
  After PS matching | 57.4 | 54.2

2. Primary Outcome: Percentage of Patients Smoking
Description: Percentage of patients with current/past smoking in the electronic medical records (EMR) are presented. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching: number analyzed (Participants) | 112 | 255
  Before PS matching | 50.0 | 51.8
  After PS matching: number analyzed (Participants) | 88 | 97
  After PS matching | 50.0 | 50.5

3. Primary Outcome: Percentage of Patients With Alcohol Consumption
Description: Percentage of patients with alcohol consumption in the electronic medical records (EMR) are presented. The patients with light to moderate, heavy and unknown quantity of alcohol consumption are considered. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching: number analyzed (Participants) | 17 | 51
  Before PS matching | 47.1 | 50.9
  After PS matching: number analyzed (Participants) | 14 | 18
  After PS matching | 50.0 | 38.9

4. Primary Outcome: Percentage of Patients With Abnormal Renal Function
Description: Percentage of patients with abnormal renal function; defined as "Any note of: Dialysis, renal transplant Serum Creatinine >1.3 Milligrams per Deciliter (mg/dL) in the electronic medical records (EMR)". Response was considered to be truly absent if not recorded in the EMR. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching | 5.5 | 11.7
  After PS matching: number analyzed (Participants) | 846 | 846
  After PS matching | 6.5 | 8.0

5. Primary Outcome: Percentage of Patients With Bleeding History or Predisposition
Description: Percentage of patients with bleeding history or predisposition is presented, defined as any note of major bleeding requiring hospitalization or blood transfusion or causing a decrease in hemoglobin level of > 2 gram per liter (g/L) in the electronic medical records (EMR). Response was considered to be truly absent if not recorded in the EMR. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching | 3.4 | 4.7
  After PS matching: number analyzed (Participants) | 846 | 846
  After PS matching | 3.7 | 4.6
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Warfarin; The concordance statistic is equal to the area under a receiver operating characteristic (ROC) curve. The C-statistic (sometimes called the "concordance" statistic or C-index) is a measure of goodness of fit for binary outcomes in a logistic regression model; Test type: Other; Regression, Logistic; Logistic regression with bleeding history or predisposition as dependent and treatment groups and claims based variables as the independent variables; C-Statistic = 0.81 — The C-statistic can be between 0.5 and 1 and a value of 0.5 indicates that the model is no better than chance at making a prediction and a value of 1.0 indicates that the model perfectly identifies those within a group and those not

6. Primary Outcome: EMR Characteristic: Renal Function - Glomerular Filtration Rate (GFR)
Description: EMR characteristic: Renal function - Glomerular Filtration Rate (GFR). Estimated GFR closest to index dispensing. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliter/minute/1.73 square meter
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Milliliter/minute/1.73 square meter
  Before PS matching: number analyzed (Participants) | 574 | 1344
  Before PS matching | 86.5 (21.6) | 78.3 (25.1)
  After PS matching: number analyzed (Participants) | 441 | 441
  After PS matching | 85.4 (21.9) | 83.4 (23.5)

7. Primary Outcome: EMR Characteristic: Serum Creatinine
Description: EMR characteristic: Serum Creatinine closest to index dispensing. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Milligrams per deciliter
  Before PS matching: number analyzed (Participants) | 574 | 1343
  Before PS matching | 1.0 (0.3) | 1.1 (0.6)
  After PS matching: number analyzed (Participants) | 441 | 441
  After PS matching | 1.0 (0.3) | 1.0 (0.4)
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Warfarin; R-squared is a statistical measure of how close the data are to the fitted regression line. 0% indicates that the model explains none of the variability of the response data around its mean. 100% indicates that the model explains all the variability of the response data around its mean; Test type: Other; Regression, Linear; Logistic regression model with serum creatinine as the dependent variable and treatment groups and claims based variables as the independent variables; Adjusted R squared statistic = 0.02 — The adjusted R² statistic, or coefficient of determination, is the proportion of the variance in the (EMR) outcome that is predictable from the independent (claims) variables, adjusted for the number of predictors in the model

8. Primary Outcome: Percentage of Patients With Abnormal Liver Function
Description: Percentage of patients with abnormal liver function; defined as "Any note of: Liver disease, cirrhosis, Active hepatitis C, Active hepatitis B, Active hepatitis A, aspartate transaminase/alanine transaminase (AST/ALT) >3 times upper limit of normal in the electronic medical records (EMR). Absence of any note would be considered as absence of the disease". Response was considered to be truly absent if not recorded in the EMR. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching | 0.5 | 0.7
  After PS matching: number analyzed (Participants) | 846 | 846
  After PS matching | 0.5 | 0.0

9. Secondary Outcome: EMR Characteristic: Duration of Atrial Fibrillation
Description: EMR characteristic: Duration of atrial fibrillation (Years / months prior to initiation of Dabigatran / Warfarin). Duration is defined as number of months prior to index date for the earliest note. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: Two sets of results are provided, before and after PS matching. Rivaroxaban and Apixaban correspond to post-hoc analyses not pre-specified in the protocol and hence not included in the outcome measures. Duration calculated for patients identified as having condition in EMR.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Months
  Before PS matching: number analyzed (Participants) | 519 | 983
  Before PS matching | 22.5 (33.8) | 26.4 (32.5)
  After PS matching: number analyzed (Participants) | 386 | 350
  After PS matching | 22.7 (35.2) | 25.4 (33.0)
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Warfarin; [analysis description as in outcome 7, analysis 1]; Test type: Other; Regression, Linear; Linear regression model with duration of atrial fibrillation as dependent and treatment groups and claims based variables as independent variables; Adjusted R squared statistic = 0.04 — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: EMR Characteristic: History of Adherence: Non-adherent/Adherent
Description: EMR characteristic: History of adherence: non-adherent/adherent.
Time Frame: Up to 12 months
Population: Two sets of results are provided, before and after PS matching. Rivaroxaban and Apixaban correspond to post-hoc analyses not pre-specified in the protocol and hence not included in the outcome measures. Although the original intent was to document the patient's history of adherence, no such information was available in the EMR
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: EMR Characteristic: History/Duration of Hypertension
Description: EMR characteristic: History/duration of hypertension. Any note of: Hypertension systolic blood pressure (SBP) >120 millimeters of mercury (mmHg) Hypertension drugs. Duration is defined as number of months prior to index date for the earliest note. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Months
  Before PS matching: number analyzed (Participants) | 938 | 2190
  Before PS matching | 42.4 (42.8) | 43.8 (41.5)
  After PS matching: number analyzed (Participants) | 708 | 726
  After PS matching | 43.6 (43.7) | 40.9 (40.6)

12. Secondary Outcome: Percentage of Patients With Uncontrolled Hypertension
Description: Percentage of patients with uncontrolled hypertension; defined as "SBP >160 mmHg using the most recent information prior to index date in the electronic medical records (EMR)". The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching: number analyzed (Participants) | 27 | 18
  Before PS matching | 0.0 | 0.0
  After PS matching: number analyzed (Participants) | 12 | 9
  After PS matching | 0.0 | 0.0

13. Secondary Outcome: EMR Characteristic: History/Duration of Congestive Heart Failure (CHF)
Description: EMR characteristic: History/duration of Congestive Heart Failure (CHF). Duration is defined as number of months prior to index date for the earliest note. Response was considered to be truly absent if not recorded in the EMR. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Months
  Before PS matching: number analyzed (Participants) | 56 | 190
  Before PS matching | 28.2 (30.8) | 38.3 (38.6)
  After PS matching: number analyzed (Participants) | 44 | 51
  After PS matching | 26.0 (30.1) | 33.9 (38.0)

14. Secondary Outcome: Percentage of Patients With Prior Transient Ischemic Attack
Description: Percentage of patients with any note of prior transient ischemic attack in the electronic medical records (EMR). Response was considered to be truly absent if not recorded in the EMR. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching | 1.6 | 2.1
  After PS matching: number analyzed (Participants) | 846 | 846
  After PS matching | 1.4 | 2.4

15. Secondary Outcome: Percentage of Patients With Diabetes
Description: Percentage of patients with any note of diabetes type I or II in the electronic medical records (EMR) is presented. Response was considered to be truly absent if not recorded in the EMR. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching | 13.4 | 18.2
  After PS matching: number analyzed (Participants) | 846 | 846
  After PS matching | 14.7 | 14.5
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Warfarin; The concordance statistic is equal to the area under a ROC curve. The C-statistic (sometimes called the "concordance" statistic or C-index) is a measure of goodness of fit for binary outcomes in a logistic regression model; Test type: Other; Regression, Logistic; Logistic regression model with diabetes as the dependent variable and treatment groups and claims based variables as the independent variables; C-Statistic = 0.88 — [estimate comment as in outcome 5, analysis 1]

16. Secondary Outcome: Percentage of Patients With Hyperlipidemia
Description: Percentage of patients with hyperlipidemia is presented, defined as any note of hyperlipidemia, dyslipidemia or Low Density Lipoprotein (LDL) >130 mg/dl in the electronic medical records (EMR). Response was considered to be truly absent if not recorded in the EMR. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching | 34.8 | 36.8
  After PS matching: number analyzed (Participants) | 846 | 846
  After PS matching | 35.6 | 34.0
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Warfarin; [analysis description as in outcome 15, analysis 1]; Test type: Other; Regression, Logistic; Logistic regression model with hyperlipidemia as the dependent variable and treatment groups and claims based variables as the independent variables; C-Statistic = 0.69 — [estimate comment as in outcome 5, analysis 1]

17. Secondary Outcome: EMR Characteristic: Hypertension, Abnormal Liver/Renal Function, Stroke, Bleeding History or Predisposition, Labile International Normalized Ratio, Elderly, Drugs/Alcohol Usage (HAS-BLED) Score
Description: EMR characteristic: HAS-BLED Score. HAS-BLED score is calculated by adding the specified points for each of the conditions listed below. Hypertension (uncontrolled), Abnormal renal and liver function, Stroke, Bleeding history or predisposition (anemia), Labile International Normalized Ratio (INR), Elderly, Drugs or alcohol (1 point each). Labile INR is defined as as the most recent INR <2 or >3 prior to cohort entry. Conditions are considered to be truly absent if not recorded in the EMR. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 12 months
Population: Two sets of results are provided, before and after PS matching. Rivaroxaban and Apixaban correspond to post-hoc analyses not pre-specified in the protocol and hence not included in the outcome measures. Also the patients with data for all HAS-BLED components.
Measure: Mean (Standard Deviation); unit: Unit on Scale
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Unit on Scale
  Before PS matching | 1.4 (1.0) | 1.6 (1.0)
  After PS matching: number analyzed (Participants) | 846 | 846
  After PS matching | 1.5 (1.0) | 1.5 (1.0)
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Warfarin; [analysis description as in outcome 7, analysis 1]; Test type: Other; Regression, Linear; Linear regression model with HAS-BLED score as the dependent variable and treatment groups and claims based variables as the independent variables; Adjusted R squared statistic = 0.34 — [estimate comment as in outcome 7, analysis 1]

18. Secondary Outcome: Percentage of Patients With Use of Antiplatelets or Non-steroidal Anti-inflammatory Drugs
Description: Percentage of patients with use of antiplatelets or non-steroidal anti-inflammatory drugs (NSAIDs). Includes use of aspirin, clopidogrel, prasugrel, ticagrelor or NSAIDs (within 1 month or on the index date) in the electronic medical records (EMR). Response was considered to be truly absent if not recorded in the EMR. The results are provided before and after propensity score (PS) matching. Before PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR whose data were available; After PS matching: all patients meeting inclusion/exclusion criteria successfully linked to EMR, 1:1 propensity score matched, whose data were available.
Time Frame: Up to 1 month
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 1130 | 2566
Percentage of patients
  Before PS matching | 18.0 | 18.4
  After PS matching: number analyzed (Participants) | 846 | 846
  After PS matching | 17.1 | 18.7

ADVERSE EVENTS:
Time Frame: Safety monitoring and safety reporting on an individual case level is not applicable.
Description: Serious and other (non-serious) adverse events were not of interest in this study and therefore were not collected or assessed as part of the study, in addition individual patient data is not available therefore adverse event data is not presented.
Arm/Group | Dabigatran Etexilate | Warfarin | Rivaroxaban | Apixaban
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT03006341/Prot_SAP_000.pdf